CLINICAL TRIAL: NCT06468995
Title: Antiviral Long Acting Drugs Landing in People Living With HIV (ALADDIN): Prospective, Double-arm, Randomized, Open-label, Implementation-effectiveness Hybrid Type III Study
Brief Title: Antiviral Long Acting Drugs Landing in People Living With HIV
Acronym: ALADDIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Castagna Antonella, Prof, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CET 166-2024
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: HIV; Antiviral Agents
Keywords: Rilpivirine; Cabotegravir; HIV; Long acting; Antiretroviral; PLWH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hospital arm (Active Comparator): CAB 600mg +RPV 900mg q2M IM administration and follow-up in hospital
  Interventions: Other: Surveys completion; Drug: Hospital administration of CAB+RPV
- Home arm (Experimental): CAB 600mg +RPV 900mg q2M IM administration and follow-up at home
  Interventions: Other: Surveys completion; Drug: Home administration of CAB+RPV

INTERVENTIONS:
Other: Surveys completion — Completion of surveys: the Feasibility of Implementation Measure (FIM), the Acceptability of Intervention Measure (AIM), the Intervention Appropriateness Measure (IAM), a Likert scale, the EQ-5D-5L questionnaire, the HIV/AIDS-Targeted Quality of Life (HAT-QoL) questionnaire and the HIV Treatment Satisfaction Questionnaire (HIVTSQ).
Drug: Home administration of CAB+RPV — Drug treatment and follow-up at home (home arm).
  Arms: Home arm
Drug: Hospital administration of CAB+RPV — Drug treatment and follow-up in hospital (hospital arm)
  Arms: Hospital arm

SUMMARY:
This is a monocentric, prospective, double-arm, randomized, open-label, implementation-effectiveness hybrid type III study aimed at comparing hospital-based and home-based administration of CAB LA + RPV LA treatment for HIV-1-infected patients.

Study participants receiving IM CAB + RPV will complete various questionnaires and scales, including FIM, AIM, IAM, EQ-5D-5L, HAT-QoL, and HIVTSQ, throughout the study. HCPs will also complete FIM, AIM, IAM, and a Likert scale.

DETAILED DESCRIPTION:
This is a monocentric, prospective, double-arm, randomized, open-label, implementation-effectiveness hybrid type III study. This means that the study will focus both on implementation and effectiveness by examination of two different settings of treatment administration (hospital-based and home-based) to identify what facilitators or barriers may improve feasibility (i.e. factors that can either help or hinder the successful implementation), appropriateness and acceptability of each strategy delivery mode in order to address the needs of PLWH followed in a large clinical center in Milan, Italy.

The study will use an implementation science approach to address the question of 'what works, where and why' by identifying factors and processes that negatively and positively affect implementation outcomes from both the patients and providers perspective.

Real-world efforts to delivering the treatment to HIV-1-infected, virologically suppressed adults in two different settings (home or hospital) will be sustained.

Two healthcare delivery pathways will be explored in this study:

1. Hospital-based setting: HIV clinic nurse will administer injections at the clinic;
2. Home-patient setting: HIV clinic nurse will administer injections at patient home.

San Raffaele Hospital has participated in the phase III trials of CAB LA + RPV LA and has already developed a large experience in treating patients with LA regimes. LA administration in out-of-hospital sites could be a safe and viable option to satisfy patient needs in terms of time to move to the hospital.

Enrolled participants will be randomized, in a ratio 1:1, to the following arms:

1. drug treatment and follow-up in hospital (hospital arm);
2. drug treatment and follow-up at home (home arm).

HCPs will also be study participants. Their insight regarding feasibility, acceptability, and appropriateness of CAB LA + RPV LA administration overall and in a home-based or a hospital-based setting will be evaluated during the study period.

Cabotegravir long-acting + rilpivirine long-acting (CAB LA + RPV LA) is a licensed new drug, already used in clinical practice, for the treatment of HIV infection.

At the discretion of the person with HIV and the physician, there are two ways to begin the long acting therapy regimen:

* By taking the two drugs cabotegravir and rilpivirine orally for about a month (one tablet each), taken together 1 time a day and on a full stomach, and then switching to injectable (LA) formulations (optional according to clinical practice).
* Directly with injectable formulation.

In this study IM CAB + RPV will be delivered in the hospital-based or the home-based setting. Injections will be delivered by HCPs in the two study settings.

Study participants living with HIV receiving IM CAB + RPV, HCPs will provide their insight on the implementation of LA IM CAB+RPV by means of questionnaires and scales over the study period.

Study participants living with HIV receiving IM CAB + RPV will be asked to complete the Feasibility of Implementation Measure (FIM), the Acceptability of Intervention Measure (AIM), the Intervention Appropriateness Measure (IAM), a Likert scale, the EQ-5D-5L questionnaire, the HIV/AIDS-Targeted Quality of Life (HAT-QoL) questionnaire and the HIV Treatment Satisfaction Questionnaire (HIVTSQ).

HCPs will be asked to complete the Feasibility of Implementation Measure (FIM), the Acceptability of Intervention Measure (AIM), the Intervention Appropriateness Measure (IAM) and a Likert scale.

Study participants receiving drug treatment will be treated in the home-based or hospital-based study setting for 12 [1 month for screening + 11 of hospital or home treatment administration, in accordance to the clinical practice. People receiving optional OLI according to clinical practice will receive oral antiretrovirals in the month before baseline. HCPs are responsible for the administration of LA IM CAB + RPV in the two study settings.

People receiving LA IM CAB + RPV in the hospital setting will receive injections as per medical practice in dedicated spaces within the Infectious Diseases Unit of San Raffaele Hospital.

People receiving LA IM CAB + RPV in the home-based setting will receive injections at their home within the Metropolitan Area of Milan. HCPs will directly reach the study participant's home. Administration of CAB + RPV, completion of study surveys, blood collection for laboratory exams according to clinical practice and all study procedures will be performed by the HCPs at the study participant home.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV-1 infection that could, according to clinical practice, switch current ART to IM CAB + RPV;
* Aged 18 years or older at the time of signing the informed consent.
* People willing to switch to long-acting therapy
* on a stable (≥6 months) antiretroviral regimen and virologically suppressed (HIV-1 RNA <50 copies/ml):

  * Documented evidence of plasma HIV-1 RNA measurements <50 c/mL in the 6 months prior to Screening.
  * Plasma HIV-1 RNA <50 c/mL at Screening.
* Ability to understand informed consent form and other relevant regulatory documents.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Within 6 months prior to Screening, any plasma HIV-1 RNA measurement >=50 c/mL or within the 6 to 12-month window prior to Screening, any plasma HIV-1 RNA measurement >200 c/mL, or 2 or more plasma HIV-1 RNA measurements >=50 c/mL.
* Present or past evidence of viral resistance to agents of the NNRTI or INI class or prior treatment failure with agents of NNRTI or INSTI class
* Unwillingness or any condition that might prevent the completion of all surveys over study follow-up.
* Any contraindication for CAB LA, RPV LA, oral Cabotegravir or Rilpivirine (see EU SmPC):

  * Women who are pregnant, breastfeeding or plan to become pregnant or breastfeed during the study
  * Any evidence of a current Center for Disease Control and Prevention (CDC) Stage 3 disease, except cutaneous Kaposi's sarcoma not requiring systemic therapy, and CD4+ counts <200 cells/mL are not exclusionary
  * Participants with moderate to severe hepatic impairment
  * Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant
  * Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV DNA as follows:

    * Participants positive for HBsAg are excluded;
    * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status), whether negative or positive for HBV DNA, are excluded
* Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.

  * Asymptomatic individuals with chronic hepatitis C virus (HCV) infection will not be excluded, however Clinicians must carefully assess if therapy specific for HCV infection is required; participants who require or qualify for immediate HCV treatment are excluded
  * Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis, or decompensated cirrhosis (eg. ascites, encephalopathy, or variceal bleeding)), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment)
  * History of liver cirrhosis with or without hepatitis viral co-infection.
  * Ongoing or clinically relevant pancreatitis
  * Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical and anal intraepithelial neoplasia.
  * History or presence of allergy or intolerance to the study drugs or their components or drugs of their class. In addition, if heparin is used during pharmacokinetic sampling, participants with a history of sensitivity to heparin or heparin-induced thrombocytopenia must not be enrolled.
  * Current platelet count<100,000 x109/L.
  * Any evidence of primary resistance based on the presence of any major known Integrase inhibitor (INI) or Non-nucleoside reverse transcriptase inhibitor (NNRTI) resistance-associated mutation, except for K103N by any historical resistance test result.
  * Any verified Grade 4 laboratory abnormality at screening.
  * Subjects has estimated creatinine clearance <50mL/minute per 1.73-meter square via Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) Method
  * Alanine aminotransferase (ALT) >=3 × Upper limit of normal (ULN)
  * Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
  * Use of medications which are associated with Torsade de Pointes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Implementation Measure (FIM) scale | Months 1 and 7 and 11
  Proportion of participants receiving injections with an average composite score greater than or equal to 4 across the questions of Feasibility of Implementation Measure (FIM) and average composite score.
Acceptability of Intervention Measure (AIM) scale | Months 1 and 7 and 11
  Proportion of participants receiving injections with an average composite score greater than or equal to 4 across the questions of Acceptability of Intervention Measure (AIM) and average composite score.
Intervention Appropriateness Measure (IAM) scale | Months 1 and 7 and 11
  Proportion of participants receiving injections with an average composite score greater than or equal to 4 across the questions of Intervention Appropriateness Measure (IAM) and average composite score.
Qualitative insights | Months 1 and 7 and 11
  Qualitative insights regarding feasibility, acceptability, and appropriateness of CAB+RPV IM q2M.

SECONDARY OUTCOMES:
Proportion of patients willing to enroll in the study | Months 7 and 11
  Proportion of patients willing to enroll in the study out of total screened to assess the uptake, and fidelity of CAB LA + RPV LA administration overall and in a home-based or hospital-based setting.
Proportion of patients voluntary asking to stop CAB+RPV LA administration | Months 7 and 11
  Proportion of patients voluntary asking to stop CAB+RPV LA administration out of total enrolled in the study to assess the uptake, and fidelity of CAB LA + RPV LA administration overall and in a home-based or hospital-based settingy
Proportion of CAB+RPV LA injections occurring within the target window | Months 7 and 11
  Proportion of CAB+RPV IM injections occurring within the target window from target date (+/- 7 days of target date) to assess the uptake, and fidelity of CAB LA + RPV LA administration overall and in a home-based or hospital-based setting
Average score of satisfaction on a Likert scale | Months 7 and 11
  Average score of satisfaction on a Likert scale for each implementation strategy used and qualitative insights into the relative value of the strategies and any adaptations informed by Consolidated Framework for Implementation Research Constructs (CFIR) to assess the satisfaction with the implementation strategies adopted, including unanticipated adaptations, facilitators and barriers to the uptake and process of CAB LA + RPV LA from the perspectives of patients, overall and in a home-based or hospital-based setting
Proportion of PWH with HIV-RNA >50 copies/mL | Months 7 and 11
  Proportion of people with confirmed HIV-RNA >50 copies/mL to monitor safety and effectiveness of CAB LA + RPV LA administration overall and in a home-based and hospital-based setting, as per clinical practice.
Time (months) to LA discontinuation | Months 7 and 11
  Time (months) to CAB+RPV LA discontinuation from enrollment to monitor safety and effectiveness of CAB LA + RPV LA administration overall and in a home-based and hospital-based setting, as per clinical practice
Adverse Events and Serious AEs | Months 7 and 11
  Proportion of people with Adverse Events and Serious AEs to monitor safety and effectiveness of CAB LA + RPV LA administration overall and in a home-based and hospital-based setting, as per clinical practice
EQ-5D-5L questionnaire | Months 1 and 7 and 11
  Average change vs baseline on the utility value derived from EQ-5D-5L questionnaire
HIV/AIDS-Targeted Quality of Life (HAT-QoL) questionnaire | Months 1 and 7 and 11
  Average change vs baseline on the utility value derived from the nine domains scores derived from the HIV/AIDS-Targeted Quality of Life (HAT-QoL) questionnaire
HIV Treatment Satisfaction Questionnaire (HIVTSQ) | Months 1 and 7 and 11
  Average change vs baseline on the utility value derived from the nine domains scores derived from the HIV Treatment Satisfaction Questionnaire (HIVTSQ)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Nozza, MD, Principal Investigator — Vita-Salute San Raffaele University; Antonella Castagna, Prof, Study Chair — Vita-Salute San Raffaele University
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy

IPD SHARING:
Plan to Share IPD: No